CLINICAL TRIAL: NCT01704833
Title: Cognitive Behavioral Therapy for Paranoia in Schizophrenia
Acronym: CBTp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0505007908
Record Dates: First submitted 2012-09-27; First posted 2012-10-11 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Paranoid Delusions
Keywords: Psychosis; Paranoia; Cognitive Behavioral Therapy; Delusions; Group Therapy
MeSH Terms: conditions — Psychotic Disorders; Paranoid Disorders; Delusions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): This group receives 15 weeks of Paranoia-Focused Cognitive Behavioral Therapy (PFCBT) in addition to standard care.
  Interventions: Behavioral: Paranoia-Focused Cognitive Behavioral Therapy (PFCBT)
- Treatment as Usual (No Intervention): This group receives standard care only.

INTERVENTIONS:
Behavioral: Paranoia-Focused Cognitive Behavioral Therapy (PFCBT) — The PFCBT is a 15-week Program that includes weekly group and individual sessions.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The main objective of this study is to determine the preliminary efficacy of Paranoia-Focused Cognitive Behavioral Therapy (PFCBT) relative to standard care in the treatment of persecutory delusions in patients diagnosed with schizophrenia or schizoaffective Disorder.

DETAILED DESCRIPTION:
Paranoia-Focused Cognitive Behavioral Therapy (PFCBT) is a manualized intervention that combines group and individual modalities to reduce paranoia-biased information-processing and social avoidance, and to increase insight and reality testing capacity.

This is a randomized controlled clinical trial. Twenty four adults ages 18-65 with the primary DSM-IV Schizophrenia and Schizoaffective disorder and drug-refractory persecutory delusions will be recruited from outpatient clinics in New York City Metropolitan area. Participants will be randomly assigned to either experimental or control group. The experimental group will receive PFCBT in addition to standard care and the control group will receive standard care alone. PFCBT will include participation in one group session and one individual therapy session weekly over the 15 weeks. The preliminary efficacy of the intervention will be evaluated using standardized measures by blind evaluators conducted at baseline, post-treatment, and at 6-months post-termination follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Met DSM IV diagnostic criteria for schizophrenia or schizoaffective disorder, confirmed by the Clinical Structural Diagnostic Interview (SCID, First et al, 1997) -Reported persistent and distressing paranoid delusion(s);
* A minimum severity score of 4 point Persecution subscale on The Positive and Negative Syndrome Scale (PANSS)
* Had an adequate trial (6 months or more) and were stabilized on antipsychotic medications (no change in psychiatric medication prescribed in the last month

Exclusion Criteria:

-Substance misuse or medical disorder identified as the primary cause of delusions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Persecution Severity at week 16 and at week 42. | Measured at baseline, at week 16, and at week 42.
  Measured by the Persecution sub-scale on Positive and Negative Syndrome Scale (PANSS).

SECONDARY OUTCOMES:
Change from Baseline in Attributional Style at week 16. | Measured at baseline and at week 16.
  Internal Personal and Situational Attributions Questionnaire.Measures attributional style (a tendency to attribute cause for negative events to situational or personal causes).
Change from Baseline in a Tendency to Jump to Conclusions at week 16. | Measured at baseline and at week 16.
  Measured by the BEADS Task. Measures a tendency to jump to conclusions when making a judgment.
Change from Baseline in Cognitive Insight at week 16. | Measured at baseline and at week 16.
  Beck Cognitive Insight Scale. Measures cognitive insight.
Change from Baseline in Dimensions of Paranoid Delusions | Measured at baseline, at week 16 and at week 42.
  Psychotic Symptom Rating Scales (PSYRATS), Delusions. Measure dimensions of delusions.

OTHER OUTCOMES:
The Working Alliance Inventory (WAI) | Measured at week 16 (post CBT).
  Used to assess the participants' perceived alliance to the therapist.
The Empathy Scale (ES) | Measured at week 16 (post CBT).
  Measures participants' perceptions of the therapist's warmth, genuineness, and empathy.
Group Cohesiveness Scale (GCS) | Measured at week 16 (post CBT).
  Measures group cohesiveness.
Changes from Baseline in Brain Circuitry at week 42. | Measured at baseline and at week 42.
  'Linguistic threat' fMRI paradigm is used to monitor brain circuitry changes associated with PFCBT.

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Landa, Psy D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States